CLINICAL TRIAL: NCT06796439
Title: Comparative Effects of Different Stretching Protocols on Performance Enhancement in Racquet Sports.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC014554 / Tooba
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Sport Injury; Sport Performance
Keywords: Static Stretching; Dynamic Stretching; Racquet Sports; Performance; Squash; Badminton
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Two groups will be formed. One group will be the static stretching group , i.e., group A which will be asked to perform the static stretching protocol which will include warm-up, the protocol and then the cool-down exercises and it will take 20 minutes.
  In Group B, the participants will be asked to perform dynamic stretching protocol which will include warm-up, the protocol and then the cool-down exercises. This protocol will take 20 minutes.
  After performance readings will be taken in the 1st, 3rd and 6th weeks and data will be compared to find out which method is more effective to improve performance in racquet sports players.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static Stretching Technique (Experimental): Participants will perform static Stretching protocols. There were no special warm-up exercises (running and skipping) after the implementation of static stretching exercises. After the general warm-up, participants would engage in a sequence of randomized static stretches including Lower back stretch, Quads stretch, Hams Stretch, Calf Stretch and Upper limb Stretches (biceps, Triceps, Arm across chest, Arm pull and head tilt, Side stretch, backward arm stretch, Pect. stretch and Towel Stretch). All stretches were done as 3 sets of 30 seconds for 20 minutes for 5 days per week and held at the point of mild discomfort. Readings will be taken after 1st, 3rd and 6th week, respectively
  Interventions: Other: Static stretching
- Dynamic Stretching Technique (Active Comparator): Participants will be divided into two groups with sample size of 52 participants in each group.
  Participants will perform Dynamic Stretching protocols. There were no special warm-up exercises (running and skipping) after the implementation of dynamic stretching exercises. Participants would engage in a sequence of randomized static stretches including Jumping Jacks, Lunges, Trunk Circles, arm swings and butt Kicks. All stretches were done as 3 sets of 30 seconds for 20mins for 5 days per week and held at the point of mild discomfort. Readings will be taken after 1st, 3rd and 6th week, respectively
  Interventions: Other: Dynamic Stretching

INTERVENTIONS:
Other: Static stretching — Participants will be divided into two groups with sample size of 52 participants in each group.
  Group 1: Participants will perform static Stretching protocols. There were no special warm-up exercises (running and skipping) after the implementation of static stretching exercises. After the general warm-up, participants would engage in a sequence of randomized static stretches including Lower back stretch, Quads stretch, Hams Stretch, Calf Stretch and Upper limb Stretches (biceps, Triceps, Arm across chest, Arm pull and head tilt, Side stretch, backward arm stretch, Pect. stretch and Towel Stretch). All stretches were done as 3 sets of 30 seconds for 20 minutes for 5 days per week and held at the point of mild discomfort. Readings will be taken after 1st, 3rd and 6th week, respectively.
  Group 2: Participants will perform Dynamic Stretching protocols. There were no special warm-up exercises (running and skipping) after the implementation of dynamic stretching exercises. Participants wou
  Arms: Static Stretching Technique
Other: Dynamic Stretching — Group 2: Participants will perform Dynamic Stretching protocols. There were no special warm-up exercises (running and skipping) after the implementation of dynamic stretching exercises. Participants would engage in a sequence of randomized static stretches including Jumping Jacks, Lunges, Trunk Circles, arm swings and butt Kicks. All stretches were done as 3 sets of 30 seconds for 20mins for 5 days per week and held at the point of mild discomfort. Readings will be taken after 1st, 3rd and 6th week, respectively.
  Arms: Dynamic Stretching Technique

SUMMARY:
This study intends to compare the effects of Static stretching Protocols with Dynamic stretching protocols on racquet sports players to find out how these protocols affect their performance.

DETAILED DESCRIPTION:
In this study, two groups will be formed to find out the effects of static and dynamic stretching protocols on racquet sports players over a course of 6 weeks. One group is given the static stretching protocol, and the other group is given the dynamic stretching protocol, and at the end of the 1st, 3rd, and 6th weeks, readings are taken to compare the effects of these techniques on the performance of the subjects enrolled in this study. A total of 52 participants will be involved, and the groups will be divided into 26, 26 each. Data will be analyzed through SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Males.
* Age 20- 40 years.
* Amateur Active players with at least 1 year of regular experience.
* Free from any musculoskeletal injuries or conditions affecting participation.
* Willing to provide written informed consent.

Exclusion Criteria:

* Players with ongoing or recent (<3 months) musculoskeletal injuries.
* Those with chronic conditions (e.g., arthritis, cardiovascular issues) affecting physical activity.
* Those suffering with any medical condition that affects their performance.
* Participants who are currently following a specialized stretching regimen outside regular squash warm-ups.
* Use of medications that could affect muscle function or perception during the Study.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-02 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Static Stretching Protocol | 6 weeks approximately after the study starts
  Two Groups will be formed. One group will be the static stretching group , i.e., group A which will be asked to perform the static stretching protocol which will include warm-up, the protocol and then the cool-down exercises and it will take 20 minutes.

SECONDARY OUTCOMES:
Dynamic Stretching Protocol | 6 weeks approximately after the study starts
  Two groups will be formed. In Group B, the participants will be asked to perform dynamic stretching protocol which will include warm-up, the protocol and then the cool-down exercises. This protocol will take 20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Riafat Mehmood, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No